CLINICAL TRIAL: NCT00623571
Title: Acute Exacerbation of Chronic Heart Failure: "Hospital at Home" Versus Inpatient Care for Elderly Patients. A Randomized, Controlled Trial.
Brief Title: Hospitalization at Home of Elderly Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 516
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2004-01

CONDITIONS: Heart Failure
Keywords: frail elderly; hospital at home; heart failure; Acute exacerbation of chronic heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients treated by hospital-at-home service (GHHS)
  Interventions: Other: Treatment of elderly patients in GHHS
- 2 (Active Comparator): Patients treated in a general medical ward (GMW)
  Interventions: Other: Treatment of elderly patients in a GMW

INTERVENTIONS:
Other: Treatment of elderly patients in a GMW
  Arms: 2
Other: Treatment of elderly patients in GHHS
  Arms: 1

SUMMARY:
Aim of the study was to evaluate the efficacy of hospital-at-home treatment compared with inpatient care in selected elderly patients with acute exacerbation of chronic heart failure (CHF).

DETAILED DESCRIPTION:
A total of 101 elderly patients admitted to the emergency department of the hospital for acute exacerbation of CHF were randomly assigned to a general medical ward (GMW, n = 53) or to a geriatric home hospitalization service (GHHS, n = 48).

All patients aged 75 and older admitted to the ED (Emergence Department) of the San Giovanni Battista Hospital during the period between April 2004 and April 2005 with main diagnosis of heart failure and requiring acute hospitalization were enrolled in the study.

Additional inclusion criteria were appropriate care supervision at home, telephone connection, living in the hospital-at-home catchment area and informed consent. Exclusion criteria were absence of family and social support; patients who need mechanical ventilation, severe dementia, end-stage cancer, history of severe renal impairment or hepatic failure with ascitis.

All patients involved underwent a baseline standard clinical evaluation, blood tests that included haematocrits, glycemia, hepatic and renal function and electrolytes, and instrumental investigations. Only those who had been evaluated in the ED for at least 12 to 24 hours were considered eligible for the study.

Patients fulfilling inclusion criteria were informed about the nature of the study and asked to give their informed consent. Extensive information was also provided to patient's relatives to obtain their collaboration.

Directly in the ED, eligible patients were randomly assigned to GHHS or to a GMW and immediately transferred. For the randomization, a set of computer-generated random numbers in a 1:1 ratio has been used. The allocation sequence was unknown to any of the investigators and was contained in a set of sealed envelopes, each bearing on the outside only the name of the hospital and a number.

Measurements of baseline sociodemographic information, clinical data, functional, cognitive and nutritional status, depression and quality of life were obtained for the entire sample.

Patients transferred home were immediately visited by members of the hospital at home's team who conducted a multidimensional geriatric assessment and programmed the home treatment that was the same that hospitalised patients received. In addition, patients treated at home and their caregivers obtained adequate education about the knowledge of the disease and constant advice about smoking cessation, nutrition, use of drugs and early recognition of triggers of disease's exacerbation. The GHHS group received a daily nurse visit and a physician's visit every two or three days for the entire length of stay. The inpatients control group received routine hospital care. Hospital at home staff was available at all times for urgent home visits.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of chronic heart failure,
* Age over 75,
* Appropriate care supervision at home,
* Telephone connection,
* Living in the hospital-at-home catchment area and informed consent.

Exclusion Criteria:

* Absence of family and social support;
* Patients who need mechanical ventilation,
* Severe dementia,
* End-stage cancer,
* History of severe renal impairment or hepatic failure with ascitis.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
mortality | 6 months

SECONDARY OUTCOMES:
hospital readmissions | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Geriatric Department of San Giovanni Battista Hospital, Torino, Torino, Italy

REFERENCES:
- [Derived] Tibaldi V, Isaia G, Scarafiotti C, Gariglio F, Zanocchi M, Bo M, Bergerone S, Ricauda NA. Hospital at home for elderly patients with acute decompensation of chronic heart failure: a prospective randomized controlled trial. Arch Intern Med. 2009 Sep 28;169(17):1569-75. doi: 10.1001/archinternmed.2009.267. PMID 19786675